CLINICAL TRIAL: NCT01246765
Title: National Pregnancy Registry for Psychiatric Medications
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Alkermes, Inc. (Industry); Eisai Inc. (Industry); Otsuka America Pharmaceutical (Industry); Supernus Pharmaceuticals, Inc. (Industry); Sage Therapeutics (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Lee S. Cohen, MD, Director, MGH Center for Women's Mental Health, Massachusetts General Hospital
Other Study IDs: 2008P-001861
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Pregnant Women; Psychotropic Drugs
Keywords: Pregnancy; Medication use during pregnancy; Psychiatric medications; ADHD; Atypical Antipsychotics; Antidepressants; Sedative Hypnotics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Atypical Antipsychotic Cohort: Pregnant women who have taken at least one type of atypical antipsychotic at some point during pregnancy.
  Medications of Special Interest:
  * Abilify (aripiprazole)
  * Aristada (aripiprazole lauroxil)
  * Aristada Initio (aripiprazole lauroxil)
  * Clozaril (clozapine)
  * Lybalvi (olanzapine and samidorphan)
  * Rexulti (brexpiprazole)
  * Risperdal (risperidone)
  * Seroquel (quetiapine)
  * Symbax (olanzapine-fluoxetine HCL)
  * Zyprexa (olanzapine)
- Antidepressant Medications: Pregnant women who have taken at least one type of antidepressant medication at some point during pregnancy.
  Medications of Special Interest:
  * Spravato (esketamine)
  * Zulresso (brexanolone)
- ADHD Medications: Pregnant women who have taken at least one type of ADHD medication at some point during pregnancy.
  Medications of Special Interest:
  • Qelbree (viloxazine)
- Sedative Hypnotic Medications: Pregnant women who have taken at least one type of sedative hypnotic medication at some point during pregnancy.
  Medications of Special Interest:
  • Dayvigo (lemborexant)
- Other Psychiatric Medications: Pregnant women who have taken other psychiatric medications (other than atypical antipsychotics, ADHD medications, antidepressants, or sedative hypnotics) at some point during pregnancy.

SUMMARY:
The National Pregnancy Registry for Psychiatric Medications is dedicated to evaluating the safety of psychiatric medications such as antidepressants, ADHD medications, sedative hypnotics, and atypical antipsychotics that many people take during pregnancy to treat a wide range of mood, anxiety, executive function, or psychiatric disorders. The goal of this Registry is to gather information on the safety of these medications during pregnancy, as current data is limited.

DETAILED DESCRIPTION:
The overarching objectives of the National Pregnancy Registry for Psychiatric Medications are twofold: to assess risk for malformations among infants exposed to specific psychiatric medications and to assess neonatal outcomes associated with prenatal exposure to such medication. Specifically, the Registry will allow us to prospectively determine whether exposure to psychiatric medication is associated with any increased risk for major malformations above the baseline risk noted in the general population. This will be achieved by careful systematic documentation of medication exposure during pregnancy, as well as other relevant exposures often not included in small case series or published reviews of drug safety derived from large administrative databases.

Although psychiatric medications are widely used by reproductive age women, reliable data regarding the reproductive safety of many of these compounds is limited. As a result, clinicians often lack sufficient evidence to evaluate the risks and benefits of using medications to treat psychiatric disorders during pregnancy. The National Pregnancy Registry for Psychiatric Medications is one of the first, and largest, hospital-based pregnancy registries which will systematically and prospectively monitor pregnancy outcomes after exposure to psychiatric medications, including antidepressants, ADHD medications, sedative hypnotics, and atypical antipsychotics.

Primary Aim:

To prospectively evaluate rates of congenital malformations among infants exposed in-utero to psychiatric medications.

Secondary Aims:

1. To evaluate neonatal outcomes of infants with prenatal exposure to specific psychiatric medications alone or in combination with other psychotropics.
2. To evaluate maternal health outcomes associated with use of psychiatric medications during pregnancy.
3. To evaluate neurobehavioral development of children (1 month and older) with prenatal exposure to psychiatric medications.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Age 18-45
* Subjects will be willing to participate over the phone
* Subjects will be able to provide informed consent

Exclusion Criteria:

* Women who have completed their pregnancy
* Women who are planning to become pregnant
* Women who are not taking any psychiatric medications and/or have no history of psychiatric illness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women from across the United States will be enrolled in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2008-11 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Major Malformations in Infants | Birth up to 1 year; assessed at 8-12 weeks postpartum, assessed through medical records through 1 year of age.
  The primary outcome for this study is rates of major malformations among infants exposed in-utero to psychiatric medications. A major malformation is defined as a structural abnormality with surgical, medical, or cosmetic importance. Exclusions include (1) minor anomalies; (2) deformations; (3) physiologic features due to prematurity, such as undescended testes; (4) birthmarks; (5) genetic disorders and chromosomal abnormalities; and (6) any finding by prenatal sonography, such as absence of 1 kidney, or at surgery (or autopsy) that was not identified by an examining pediatrician. This data is collected through review of pediatric medical records through the first twelve months of infants' lives.

SECONDARY OUTCOMES:
Maternal Gestational Weight Gain | Change from pre-pregnancy to delivery; assessed at 7 months' gestation and 8-12 weeks postpartum.
  Maternal gestational weight gain is measured by the change in maternal weight from pre-pregnancy to weight at delivery, recorded in pounds.
Live Birth | Birth; assessed at 8-12 weeks postpartum.
  Did the pregnancy end in a live birth, assessed as a yes/no outcome.
Spontaneous Abortion (SAB) | Any time during pregnancy; assessed at 7 months' gestation and 8-12 weeks postpartum.
  Did a spontaneous abortion (SAB) occur during the pregnancy, assessed as a yes/no outcome.
Intrauterine Fetal Demise (IUFD) | Any time during pregnancy; assessed at 7 months' gestation and 8-12 weeks postpartum.
  Did intrauterine fetal demise (IUFD) occur during the pregnancy, assessed as a yes/no outcome.
Gestational Age | Birth; assessed at 8-12 weeks postpartum.
  The gestational age of the infant at birth, recorded in weeks and days.
Preterm Delivery | Any time during pregnancy; assessed at 7 months' gestation and 8-12 weeks postpartum.
  Was the baby born before 37 weeks gestational age, assessed as a yes/no outcome.
Birth Weight | Birth; assessed at 8-12 weeks postpartum.
  Birth weight of the infant, recorded in grams or lbs and oz
Delivery Method | Birth; assessed at 8-12 weeks postpartum.
  Was birth vaginal or by C-section; if C-section, emergent: yes/no
Gestational Diabetes | Any time during pregnancy; assessed at baseline, 7 months' gestation and 8-12 weeks postpartum.
  Gestational diabetes diagnosed during pregnancy, assessed as a yes/no outcome.
Gestational Hypertension | Any time during pregnancy; assessed at baseline, 7 months' gestation and 8-12 weeks postpartum.
  Gestational hypertension diagnosed during pregnancy, assessed as a yes/no outcome.
Preeclampsia/Eclampsia | Any time during pregnancy; assessed at baseline, 7 months' gestation and 8-12 weeks postpartum.
  Pre-eclampsia or eclampsia diagnosed during pregnancy, assessed as a yes/no outcome.
Maternal Postpartum Hemorrhage | Birth; assessed at 8-12 weeks postpartum.
  Did maternal postpartum hemorrhage occur, assessed as a yes/no outcome.
Apgar Scores | Birth; assessed at 8-12 weeks postpartum.
  1-min and 5-min Apgar scores.
Neonatal Intensive Care Unit (NICU) admission | Birth up to 1 year; assessed at 8-12 weeks postpartum, assessed through medical records through 1 year of age.
  Was the infant admitted to the NICU, assessed as a yes/no outcome; if yes, number of days in NICU and reason for admission
Infant Death | Birth up to 1 year; assessed at 8-12 weeks postpartum, assessed through medical records through 1 year of age.
  Did the infant die before the age of one; assessed as a yes/no outcome.
Neonatal Extrapyramidal Symptoms | Birth through 1 year; assessed at 8-12 weeks postpartum, assessed through medical records through 1 year of age.
  Did movement dysfunction occur in the infant (such as dystonia, akathisia, parkinsonism characteristic symptoms such as rigidity, bradykinesia, tremor, and tardive dyskinesia); assessed as a yes/no outcome.
Poor Neonatal Adaptation Syndrome (PNAS) | Birth through 1 year; assessed at 8-12 weeks postpartum, assessed through medical records through 1 year of age.
  Did poor neonatal adaptation syndrome (PNAS) occur (including poor muscle tone, tremors, jitteriness, irritability, seizures, feeding difficulties, sleep disturbances, hypoglycemia, and respiratory distress); assessed as a yes/no outcome
Child Development Outcomes - Ages and Stages Questionnaire (ASQ-3) | Assessed at 9 months, year 3, and year 5.
  Were there developmental concerns, as assessed by the Ages and Stages Questionnaire (ASQ-3).
Child Development Outcomes - Preschool Child Behavior Checklist (CBCL) | Assessed at 9 months, year 3, and year 5.
  Were there developmental concerns, as assessed by the Preschool Child Behavior Checklist (CBCL).
Breastfeeding | Assessed at 8-12 weeks postpartum.
  Did breastfeeding occur, assessed as a yes/no outcome; if yes, duration of breastfeeding recorded in weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Cohen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen LS, Viguera AC, McInerney KA, Freeman MP, Sosinsky AZ, Moustafa D, Marfurt SP, Kwiatkowski MA, Murphy SK, Farrell AM, Chitayat D, Hernandez-Diaz S. Reproductive Safety of Second-Generation Antipsychotics: Current Data From the Massachusetts General Hospital National Pregnancy Registry for Atypical Antipsychotics. Am J Psychiatry. 2016 Mar 1;173(3):263-70. doi: 10.1176/appi.ajp.2015.15040506. Epub 2015 Oct 6. PMID 26441156
- [Derived] Swetlik C, Cohen LS, Kobylski LA, Sojka ET, Killenberg PC, Freeman MP, Viguera AC. Effects of Prenatal Exposure to Second-Generation Antipsychotics on Development and Behavior Among Preschool-Aged Children: Preliminary Results From the National Pregnancy Registry for Psychiatric Medications. J Clin Psychiatry. 2024 Mar 13;85(1):23m14965. doi: 10.4088/JCP.23m14965. PMID 38488388
- [Derived] Szpunar MJ, Freeman MP, Kobylski LA, Rossa ET, Gaccione P, Chitayat D, Viguera AC, Cohen LS. Risk of Major Malformations in Infants After First-Trimester Exposure to Stimulants: Results From the Massachusetts General Hospital National Pregnancy Registry for Psychiatric Medications. J Clin Psychopharmacol. 2023 Jul-Aug 01;43(4):326-332. doi: 10.1097/JCP.0000000000001702. Epub 2023 May 29. PMID 37235505
- [Derived] Viguera AC, Freeman MP, Kobylski LA, Rossa ET, Gaccione P, Chitayat D, Hernandez-Diaz S, Cohen LS. Risk of Major Malformations Following First-Trimester Exposure to Olanzapine: Preliminary Data From the Massachusetts General Hospital National Pregnancy Registry for Psychiatric Medications. J Clin Psychopharmacol. 2023 Mar-Apr 01;43(2):106-112. doi: 10.1097/JCP.0000000000001665. PMID 36825887
- [Derived] Cohen LS, Church TR, Freeman MP, Gaccione P, Caplin PS, Kobylski LA, Arakelian M, Rossa ET, Chitayat D, Hernandez-Diaz S, Viguera AC. Reproductive Safety of Lurasidone and Quetiapine: Update from the National Pregnancy Registry for Psychiatric Medications. J Womens Health (Larchmt). 2023 Apr;32(4):452-462. doi: 10.1089/jwh.2022.0310. Epub 2023 Jan 30. PMID 36716275
- [Derived] Viguera AC, McElheny SA, Caplin PS, Kobylski LA, Rossa ET, Young AV, Gaccione P, Goez-Mogollon L, Freeman MP, Cohen LS. Risk of Poor Neonatal Adaptation Syndrome Among Infants Exposed to Second-Generation Atypical Antipsychotics Compared to Antidepressants: Results From the National Pregnancy Registry for Psychiatric Medications. J Clin Psychiatry. 2023 Jan 4;84(1):22m14492. doi: 10.4088/JCP.22m14492. PMID 36602927
- [Derived] Szpunar MJ, Freeman MP, Kobylski LA, Caplin PS, Gaccione P, Viguera AC, Chitayat D, Hernandez-Diaz S, Cohen LS. Risk of major malformations in infants after first-trimester exposure to benzodiazepines: Results from the Massachusetts General Hospital National Pregnancy Registry for Psychiatric Medications. Depress Anxiety. 2022 Dec;39(12):751-759. doi: 10.1002/da.23280. Epub 2022 Jul 31. PMID 35909254
- [Derived] Viguera AC, Freeman MP, Goez-Mogollon L, Sosinsky AZ, McElheny SA, Church TR, Young AV, Caplin PS, Chitayat D, Hernandez-Diaz S, Cohen LS. Reproductive Safety of Second-Generation Antipsychotics: Updated Data From the Massachusetts General Hospital National Pregnancy Registry for Atypical Antipsychotics. J Clin Psychiatry. 2021 Aug 3;82(4):20m13745. doi: 10.4088/JCP.20m13745. PMID 34352165
- [Derived] Freeman MP, Viguera AC, Goez-Mogollon L, Young AV, Caplin PS, McElheny SA, Church TR, Chitayat D, Hernandez-Diaz S, Cohen LS. Reproductive safety of aripiprazole: data from the Massachusetts General Hospital National Pregnancy Registry for Atypical Antipsychotics. Arch Womens Ment Health. 2021 Aug;24(4):659-667. doi: 10.1007/s00737-021-01115-6. Epub 2021 Mar 12. PMID 33710399
- [Derived] Cohen LS, Goez-Mogollon L, Sosinsky AZ, Savella GM, Viguera AC, Chitayat D, Hernandez-Diaz S, Freeman MP. Risk of Major Malformations in Infants Following First-Trimester Exposure to Quetiapine. Am J Psychiatry. 2018 Dec 1;175(12):1225-1231. doi: 10.1176/appi.ajp.2018.18010098. Epub 2018 Aug 16. PMID 30111186
- [Derived] Panchaud A, Hernandez-Diaz S, Freeman MP, Viguera AC, MacDonald SC, Sosinsky AZ, Cohen LS. Use of atypical antipsychotics in pregnancy and maternal gestational diabetes. J Psychiatr Res. 2017 Dec;95:84-90. doi: 10.1016/j.jpsychires.2017.07.025. Epub 2017 Jul 29. PMID 28810177
- [Derived] Cohen LS, Viguera AC, McInerney KA, Kwiatkowski MA, Murphy SK, Lemon EL, Hernandez-Diaz S. Establishment of the National Pregnancy Registry for Atypical Antipsychotics. J Clin Psychiatry. 2015 Jul;76(7):986-9. doi: 10.4088/JCP.14br09418. PMID 25939066
- See also: National Pregnancy Registry for Atypical Antipsychotics Website — https://womensmentalhealth.org/research/pregnancyregistry/